CLINICAL TRIAL: NCT00722904
Title: Evaluation of Vascular Pathology With 3D, Time-Resolved Phase Contrast MRI
Brief Title: Evaluation of Vascular Pathology With 3D, Time-Resolved Phase Contrast Magnetic Resonance Imaging (MRI)
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H627-30777; H627-30777-01A
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: post-intervention surveillance of aortic coarctation; MRA and 2D phase contrast imaging; 4D Flow velocity mapping; Patients undergoing routine post-intervention surveillance of aortic coarctation; Healthy volunteers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: patients undergoing routine post-intervention surveillance of aortic coarctation
- 2: Healthy volunteers

SUMMARY:
Aortic coarctation is a relatively common cardiovascular condition with high associated mortality if not treated. Even with successful repair, however, close follow up is needed as late complications can result in significant cardiovascular morbidity. MRI, with is ability to provide both anatomic and hemodynamic information, is becoming the imaging option of choice for post-intervention surveillance. Time-resolved, three-dimensional phase contrast magnetic resonance velocity (4D Flow) profiling enables the acquisition of multidirectional blood velocity data. The technique is well suited for evaluation of blood flow patterns in the thoracic aorta. By comparing aortic flow patterns in patients status post coarctation repair with those of healthy volunteers using 4D Flow, this study intends to characterize abnormal flow patterns in these patients with the eventual goal of better understanding and predicting late complications so that preemptive intervention may be taken.

Given the potential use of 4D Flow for evaluation of other types of vascular pathology in the aorta and other vascular regions, we hope to investigate the use of the technique on a limited basis for a broader population of adult patients. Other research groups have had success evaluating peripheral stenoses, as well as intracardiac and intracranial blood flow patterns with 4D Flow.

ELIGIBILITY:
Inclusion Criteria:

Patients: primarily status post intervention for repair of aortic coarctation and undergoing routine MRI follow up, but also adult patients with other vascular pathologies undergoing routine MRI evaluation, who may be good candidates for 4D Flow blood flow analysis.

Healthy subjects: healthy members of the radiology residency program and staff at UCSF.

Exclusion Criteria:

Anyone else.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients: primarily status post intervention for repair of aortic coarctation and undergoing routine MRI follow up, but also adult patients with other vascular pathologies undergoing routine MRI evaluation, who may be good candidates for 4D Flow blood flow analysis.
  Healthy subjects: healthy members of the radiology residency program and staff at UCSF.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
predicting late complications in patients status post coarctation repair so that preemptive intervention may be taken | For at least three years following the completion of the study, the database of patients will be updated for clinically relevant information

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Higgins, MD, Principal Investigator — UCSF Department of Radiology
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Markl M, Draney MT, Hope MD, Levin JM, Chan FP, Alley MT, Pelc NJ, Herfkens RJ. Time-resolved 3-dimensional velocity mapping in the thoracic aorta: visualization of 3-directional blood flow patterns in healthy volunteers and patients. J Comput Assist Tomogr. 2004 Jul-Aug;28(4):459-68. doi: 10.1097/00004728-200407000-00005. PMID 15232376
- [Background] Hope MD, Levin JM, Markl M, Draney MT, Alley M, Herfkens RJ. Images in cardiovascular medicine. Four-dimensional magnetic resonance velocity mapping in a healthy volunteer with pseudocoarctation of the thoracic aorta. Circulation. 2004 Jun 29;109(25):3221-2. doi: 10.1161/01.CIR.0000134277.42512.D5. No abstract available. PMID 15226232
- [Background] Hope MD, Levin JM, Markl M, Draney MT, Wilson N, Herfkens RJ. 4D Magnetic Resonance Velocity Mapping: Velocity Profile of Blood-Flow Through the Thoracic Aorta in 10 Healthy Volunteers. Abstract. ISMRM 12th Scientific Meeting, 2004
- [Background] Hope MD, Levin JM, Markl M, Draney MT, Alley MT, Dunn WN, Pelc NJ, Herfkens RJ. Four-Dimensional Magnetic Resonance Velocity Mapping: Velocity Profile of Blood Flow Through the Thoracic Aorta in 10 Healthy Volunteers. Lauterbur Award. Young Investigator Research Abstract Awards, SCBT/MR, 2004.
- [Background] Shih MC, Tholpady A, Kramer CM, Sydnor MK, Hagspiel KD. Surgical and endovascular repair of aortic coarctation: normal findings and appearance of complications on CT angiography and MR angiography. AJR Am J Roentgenol. 2006 Sep;187(3):W302-12. doi: 10.2214/AJR.05.0424. PMID 16928909
- [Background] Celermajer DS, Greaves K. Survivors of coarctation repair: fixed but not cured. Heart. 2002 Aug;88(2):113-4. doi: 10.1136/heart.88.2.113. PMID 12117824
- [Background] Toro-Salazar OH, Steinberger J, Thomas W, Rocchini AP, Carpenter B, Moller JH. Long-term follow-up of patients after coarctation of the aorta repair. Am J Cardiol. 2002 Mar 1;89(5):541-7. doi: 10.1016/s0002-9149(01)02293-7. PMID 11867038
- [Background] Klipstein RH, Firmin DN, Underwood SR, Rees RS, Longmore DB. Blood flow patterns in the human aorta studied by magnetic resonance. Br Heart J. 1987 Oct;58(4):316-23. doi: 10.1136/hrt.58.4.316. PMID 3676019
- [Background] Bogren HG, Klipstein RH, Firmin DN, Mohiaddin RH, Underwood SR, Rees RS, Longmore DB. Quantitation of antegrade and retrograde blood flow in the human aorta by magnetic resonance velocity mapping. Am Heart J. 1989 Jun;117(6):1214-22. doi: 10.1016/0002-8703(89)90399-2. PMID 2729051
- [Background] Kilner PJ, Yang GZ, Mohiaddin RH, Firmin DN, Longmore DB. Helical and retrograde secondary flow patterns in the aortic arch studied by three-directional magnetic resonance velocity mapping. Circulation. 1993 Nov;88(5 Pt 1):2235-47. doi: 10.1161/01.cir.88.5.2235. PMID 8222118
- [Background] Hope TA, Markl M, Wigstrom L, Alley MT, Miller DC, Herfkens RJ. Comparison of flow patterns in ascending aortic aneurysms and volunteers using four-dimensional magnetic resonance velocity mapping. J Magn Reson Imaging. 2007 Dec;26(6):1471-9. doi: 10.1002/jmri.21082. PMID 17968892
- [Background] Saeed M, Henk CB, Weber O, Martin A, Wilson M, Shunk K, Saloner D, Higgins CB. Delivery and assessment of endovascular stents to repair aortic coarctation using MR and X-ray imaging. J Magn Reson Imaging. 2006 Aug;24(2):371-8. doi: 10.1002/jmri.20631. PMID 16786568
- [Background] Pujadas S, Reddy GP, Weber O, Tan C, Moore P, Higgins CB. Phase contrast MR imaging to measure changes in collateral blood flow after stenting of recurrent aortic coarctation: initial experience. J Magn Reson Imaging. 2006 Jul;24(1):72-6. doi: 10.1002/jmri.20613. PMID 16755530
- [Background] Frydrychowicz A, Winterer JT, Zaitsev M, Jung B, Hennig J, Langer M, Markl M. Visualization of iliac and proximal femoral artery hemodynamics using time-resolved 3D phase contrast MRI at 3T. jMRI 2007 vol. 25 pp. 1085-92. 15. Bammer R, Hope TA, Aksoy M, Alley MT. Time-resolved 3D quantitative flow MRI of the major intracranial vessels: initial experience and comparative evaluation at 1.5T and 3.0T in combination with parallel imaging. MRM 2007: 57:127-40.
- [Background] Wigstrom L, Ebbers T, Fyrenius A, Karlsson M, Engvall J, Wranne B, Bolger AF. Particle trace visualization of intracardiac flow using time-resolved 3D phase contrast MRI. Magn Reson Med. 1999 Apr;41(4):793-9. doi: 10.1002/(sici)1522-2594(199904)41:43.0.co;2-2. PMID 10332856